CLINICAL TRIAL: NCT01260337
Title: The Effects of a Pre-packaged, Portion Controlled Meal Plan on Type 2 Diabetes and Glycemic Control: A Comparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Nutrisystem, Inc. (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12987
Record Dates: First submitted 2010-09-21; First posted 2010-12-15 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2010-09

CONDITIONS: Obesity
Keywords: Weight loss; Type 2 Diabetes; Behavior Modification; portion control
MeSH Terms: conditions — Obesity; Weight Loss; Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes Support and Education (DSE) (Active Comparator)
  Interventions: Other: Diabetes Support and Education
- Portion controlled diet (PCD) (Experimental): behavior modification
  Interventions: Behavioral: Portion controlled diet

INTERVENTIONS:
Behavioral: Portion controlled diet — Participants learn skills for changing nutritional and lifestyle habits and diabetes management follow a program that includes eating a pre-packaged, portion controlled meal for weight loss in addition to attending the behavior modification groups
  Other Names: PCD
  Arms: Portion controlled diet (PCD)
Other: Diabetes Support and Education — The DSE groups will consist of educational sessions offered for diabetes support and education which will include sessions on diet/nutrition, exercise, foot care and living with diabetes.
  Other Names: DSE
  Arms: Diabetes Support and Education (DSE)

SUMMARY:
The purpose of this research study to find out whether a pre-packaged, portion controlled diet with a group behavior modification program or group diabetes support and education, is a safe and effective way for people with type 2 diabetes to lose weight and manage their diabetes.

DETAILED DESCRIPTION:
Eligible volunteers are randomly assigned to a treatment group consisting of a pre-packaged, portion controlled meal plan plus a group behavior modification program or to a control group that consists of a group diabetes support and education (DSE) program. Random assignment will be stratified by whether or not a subject is taking insulin at baseline, which will be included as a covariate in all subsequent analyses. Treatment assignments are unmasked. At the end of 24 weeks both groups will have completed 9 group sessions (weeks 0, 1, 2, 4, 8, 12, 16, 20 and 24). At week 16, each participant will meet individually with the study physician to review their progress to date. These meetings will take place at the week 16 group visit. The PCD program is aimed at achieving and maintaining a decrease in weight and providing a group behavior modification program from 0-24 weeks. The DSE program is aimed at providing diabetes support and education from weeks 0-24. A Certified Diabetes Educator (CDE) will review the effects of diet and weight loss, exercise, and medications on blood glucose levels among all participants at the individual session before any changes in dietary intake or exercise are prescribed. Participants will be counseled on strategies to prevent hypoglycemia and will be given a blood glucose meter and strips and instructed to measure their blood glucose at least two times per day while participating in the study. In addition, the causes, symptoms and treatment of hypoglycemia will be reviewed including when to contact their health care provider.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic men and non-pregnant or non-lactating women between the ages of 21 to 75
2. BMI ≥ 25 and ≤ 50
3. Subjects must be willing to comply with all study-related procedures
4. Participant with screening HbA1C ≥ 6.5 and <12.0.

Exclusion Criteria:

1. Use of Byetta (exenatide) or Symlin (pramlintide acetate) for diabetic control< 6 months. Participants must be stable on all other medications for at least 3 months for inclusion. If a participant is on a medication for less than 3 months and the study physician determines the medications will not affect the study outcomes (weight, glycemic control, etc), they can be enrolled (excluding hypertension or cholesterol medications).
2. BMI ≤24.9 or ≥ 50.1
3. Participation in another formal weight loss program within last 6 months
4. Weight loss > 5 kg during the last 6 months
5. Participation in Diabetes Support and Education Program or other formal diabetes education program within last 6 months
6. Uncontrolled hypertension (systolic blood pressure > 180 or diastolic blood pressure > 100 mmHg). Participants on medication treating hypertension for at least three months are allowable.
7. Known atherosclerotic cardiovascular disease
8. History of congestive heart failure
9. History of a non-skin malignancy within the previous 5 years
10. Any major active rheumatologic, pulmonary, hepatic, renal, dermatologic disease or inflammatory condition
11. History of testing HIV positive
12. History of alcohol or drug abuse
13. Weight-loss inducing medications or dietary supplements within 3 months prior to enrollment.
14. Participation in any weight loss study or investigational drug study within 6 weeks prior to the screening
15. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
16. Participants taking anti-depressants (SSRI's are allowed except for bupropion [Wellbutrin]) , mood stabilizers, anti-psychotics, and psychiatric medications treating any mood, psychological or psychiatric condition. Refer to Appendix 1 for medication exclusion list.
17. Participants with screening triglycerides above 500 mg
18. Uncontrolled Dyslipidemia as defined by screening LDL cholesterol of ≥ 160 mg/dL. Participants on medication treating dyslipidemia for at least 3 months are allowable.
19. Any female who tests positive on a urine pregnancy test or who reports being pregnant at screening
20. Gastrointestinal Disorders (gallbladder disease, Crohn's disease, Irritable bowel syndrome, and any GI disease that affects malabsorption).
21. An allergy to certain foods that cannot be avoided due to the nature of the packaged foods such as, but not limited to nuts, dairy, gluten, etc.
22. Non-medical related dietary restrictions, such as vegetarians
23. Neuropathy that interferes with exercise.
24. Smoking or tobacco use
25. Previous weight loss surgery.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in weight at 3 and 6 months | Baseline, 3 & 6 months
  Assess the effects of a pre-packaged, portion controlled meal plan on weight loss in overweight and obese patients with type 2 diabetes.

SECONDARY OUTCOMES:
Change in HbA1C at 3 and 6 months | Baseline, 3 & 6 Month
  Assess the effects of a pre-packaged, portion controlled meal plan on glycemic control in overweight and obese patients with type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University, Center for Obesity Research and Education
Locations (2):
- United States (2):
  - University of Pennsylvania, Center for Weight and Eating Disorders, Philadelphia, Pennsylvania
  - Temple University, The Center for Obesity Research and Education, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Foster GD, Borradaile KE, Vander Veur SS, Leh Shantz K, Dilks RJ, Goldbacher EM, Oliver TL, Lagrotte CA, Homko C, Satz W. The effects of a commercially available weight loss program among obese patients with type 2 diabetes: a randomized study. Postgrad Med. 2009 Sep;121(5):113-8. doi: 10.3810/pgm.2009.09.2046. PMID 19820280
- See also: Center for Weight and Eating Disorders — http://www.med.upenn.edu/weight/research.shtml